CLINICAL TRIAL: NCT06466993
Title: Influence on Performance of Relaxing Breathing During Rotation Pause Before Each Station of an Objective Structured Clinical Examination for Fifth Year Medical Students
Brief Title: Influence of Relaxing Breathing Before Each Station of an Objective Structured Clinical Examination
Acronym: ZENECOS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Claude Bernard University (Other)
Responsible Party: Principal Investigator, Lilot Marc, Principal Investigator, Claude Bernard University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: ZENECOS
Record Dates: First submitted 2024-06-14; First posted 2024-06-20 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Performance Anxiety; Stress; Coping Skills

STUDY DESIGN:
Intervention Model Description: Prospective randomized controlle monocentric
Who Masked: Investigator, Outcomes Assessor
Masking Description: Evaluators of performance are blind to randomisation such as outcome assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Relaxing breathing occuring during rotation of OSCE station
  Interventions: Behavioral: Intervention of standardized relaxing breathing
- Control (Active Comparator): Free time during rotation of OSCE station
  Interventions: Behavioral: Intervention of standardized relaxing breathing

INTERVENTIONS:
Behavioral: Intervention of standardized relaxing breathing — Relaxing breathing standardized to 6 respiratory cycles per minute that occur during rotation time before next station of OSCE start

SUMMARY:
SObjective and Structured Clinical Examinations (OSCEs) has been incorporated recently in the certification process as a final national undergraduate ranking examination. This exam is an additional major stressor for medical students.

The aim of this study was to compare the efficiency on stress reduction of a standardized relaxing breathing occuring during rotation of the OSCE stations just before the start of the next upcoming OSCE station, in medical student, during the OSCE.

DETAILED DESCRIPTION:
Stress generated during the curriculum might have deleterious effects on the wellbeing and the health of medical students. Objective and Structured Clinical Examinations (OSCEs) has been incorporated recently in the certification process as a final national undergraduate ranking examination. This exam is an additional major stressor for medical students.

Stress coping strategies could be implemented to help them better prepare for this examination. The aim of this study was to compare the efficiency on stress reduction of a standardized relaxing breathing as a coping interventions occuring during rotation of the OSCE stations just before the start of the next upcoming OSCE station, in medical student, during the OSCE.

ELIGIBILITY:
Inclusion Criteria:

* all volontary medical students of the second cycle that came for their exam during the sessions of June 2024 from the University of Lyon (Medecine ESt)

Exclusion Criteria:

* no exclusion criteria

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-09-05 (Estimated); Primary Completion 2024-12-17 (Estimated); Study Completion 2024-12-17 (Estimated)

PRIMARY OUTCOMES:
PERFORMANCE | obtained seven days after the objectif structured clinical examination
  Score at the objectif structured clinical examination exam from 0 minimum to 200 points maximum

SECONDARY OUTCOMES:
Mean Difference of Inner Resource | Two times : 10 minutes before objectif structured clinical examination (before training of intervention) and just 2 minutes after training of the intervention)
  Numerical Visual analog score on inner resource available perceived (from 0 to 100 : maximum)
Mean difference of perceived impact of the intervention on performance | Just five minutes after the objectif structured clinical examination
  Numerical Visual analog scales on perceived impact of the intervention on performance (from zero: negative to 100: positive)

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Rode, MD PhD, Study Chair — Lyon Est Medical Center Lyon 1 University; Evan Gouy, MD, Principal Investigator — Lyon Est Medical Center Lyon 1 University; Marion Cortet, MD PhD, Study Director — Lyon Est Medical Center Lyon 1 University

IPD SHARING:
Plan to Share IPD: No